CLINICAL TRIAL: NCT01123798
Title: The Use of Near Infrared Spectroscopy in the Diagnosis of Acute Compartment Syndrome in Injured Soldiers
Status: Completed | Type: Observational
Sponsor: J&M Shuler (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency); Somanetics Corporation (Industry)
Responsible Party: Brett Freedman, MAJ MC (MD), Landstuhl Regional Medical Center
Other Study IDs: DR080018-01
Record Dates: First submitted 2010-02-17; First posted 2010-05-14 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Acute Compartment Syndrome
Keywords: near infrared spectroscopy; lower extremity injury
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Stable controls: Uninjured soldiers to provide normative data for stable physiological status
  Interventions: Device: near-infrared spectroscopy
- Critical controls: Critically injured soldiers with no lower extremity traumatic injuries (excepting skin abrasions and small/superficial fragmentation wounds) to provide normative data for the "shock" physiological status.
  Interventions: Device: near-infrared spectroscopy
- Lower extremity trauma: Soldiers with severe traumatic lower extremity injuries in stable and shock physiologic status. This is the investigational cohort.
  Interventions: Device: near-infrared spectroscopy

INTERVENTIONS:
Device: near-infrared spectroscopy — Non-invasive monitoring device applied on the surface of the skin that emits harmless red light to measure tissue perfusion.

SUMMARY:
The purpose of this study is to define the reliability and accuracy of Near Infrared Spectroscopy (NIRS) in the detection of intra-compartmental tissue perfusion in injured and noninjured extremities over time. The investigators hypothesize that this technology, combined with vital signs, intracompartmental pressures and clinical examinations, will be useful in diagnosing acute compartment syndrome (ACS), monitoring patients at risk for ACS, and evaluating the adequacy of fasciotomy in patients treated for ACS.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* male or female
* active duty servicemen who have been evacuated from OIF or OEF through LRMC

Exclusion Criteria:

* patients not willing to provide consent
* patients in whom application of NIRS monitoring is viewed as an impediment to casualty care

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active duty OIF/OEF military personnel who have been air evacuated from theater to Landstuhl Regional Medical Center (LRMC). Ambulatory, self-care volunteers from the LRMC outpatient spine center will be identified to serve as controls for Cohort 1.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
NIRS values in various physiologic states (stable control, critically injured control, lower extremity injury) | 24-48 hours from hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Brett Freedman, MD, Principal Investigator — Landstuhl Regional Medical Center
Locations (1):
- Landstuhl Regional Medical Center, Landstuhl, Germany